CLINICAL TRIAL: NCT04253977
Title: Promoting Healthy Weight Across the Pregnancy and Postpartum Period Through Dissemination of an Evidence Based Intervention
Brief Title: Promoting Healthy Weight Across the Pregnancy and Postpartum Period
Acronym: HEALTH-P2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201909155
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Healthy Eating & Active Living Taught at Home during Pregnancy and Postpartum (HEALTH-P2) embeds content related to healthy eating and activity within Parents as Teachers (PAT)'s existing home visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEALTH-P2 (Experimental): Along with PAT National Center, parent educators affiliated with PAT sites in HEALTH-P2; with be trained to use the HEALTH-P2 training curriculum (implementation strategy).
  Interventions: Behavioral: HEALTH-P2
- Usual Care (Active Comparator): Participants at usual care PAT sites will receive PAT as usual.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: HEALTH-P2 — The HEALTH-P2 curriculum includes evidence based lifestyle change strategies to prevent excess gestational weight gain and postpartum weight retention embedded within and delivered as part of home visits.
  Arms: HEALTH-P2
Behavioral: Usual Care — The Foundational (usual care) curriculum uses a strength-based, solution-focused model to provide parents with child development knowledge and parenting support, empowering parents as their child's first and most influential teacher.
  Arms: Usual Care

SUMMARY:
This project evaluates the effectiveness of an evidence-based intervention (HEALTH-P2) to prevent excessive weight gain from pregnancy through 12 months postpartum when disseminated and implemented in real-world settings, through Parents as Teachers. To enhance the impact of HEALTH-P2, the study also evaluates implementation outcomes from the training curriculum (implementation strategy) and external validity when HEALTH-P2 is implemented within this national home visiting organization. This partnership has potential for significant impact on obesity and chronic diseases such as cardiovascular disease and diabetes.

DETAILED DESCRIPTION:
Women are exceptionally vulnerable during childbearing years to gain disproportionally large amounts of weight when compared to men or other life periods. Weight gained during pregnancy and retained after the postpartum period contributes to obesity development and progression. Evidence based lifestyle interventions addressing the trajectory of weight gain across the childbearing continuum can reverse these alarming trends of excessive weight among young women, but have had limited uptake due to time, expense, and parenting priorities. To address this gap, our research team developed the lifestyle intervention Healthy Eating, Activity Living, Taught at Home during Pregnancy and Postpartum (HEALTH-P2) in partnership with Parents as Teachers (PAT). This study will provide evidence for the dissemination and implementation (D&I) of HEALTH-P2 across PAT's network of sites, promoting healthy weight on a national scale. The study builds on our previous work with a pragmatic cluster randomized controlled trial to evaluate D&I of HEALTH-P2 across multiple levels to achieve widespread impact. First, we will determine weight outcomes (12-month postpartum weight; gestational weigh gain) among 336 overweight/obese women (N=168 HEALTH-P2; N=168 usual care) when parent educators (~8/site) from PAT sites nationwide receive the HEALTH-P2 training through PAT National Center's existing training infrastructure and conduct HEALTH-P2 as part of routine practice. From a D&I perspective, an evaluation guided by RE-AIM will measure implementation outcomes (acceptability, appropriateness, feasibility, fidelity, adaptation). Further, the Conceptual Framework for Implementation Research will guide an assessment of contextual factors that influence external validity at multiple levels (mother, parent educator, PAT site).

ELIGIBILITY:
For Parent educators:

Inclusion Criteria:

* Deliver PAT at a site participating in the study
* Provide informed consent

Exclusion Criteria:

• At least 18 years of age

For the participants:

Inclusion Criteria:

* 18-45 years of age
* pregnant
* overweight or obese (BMI over 25 kg/m2) before becoming pregnant
* English or Spanish speaking
* participating or willing to participate in PAT at a participating PAT site until baby turns 1
* able to give informed consent for participation

Exclusion Criteria:

* planning to become pregnant again before their baby turns 1
* unable to engage in a walking program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — For the participants (i.e., not the parent educators), only women will be included: Including only female participants is scientifically justified, as the study focus is addressing the gestational weight gain.
Enrollment: 784 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in weight | 12 months postpartum
  Mother's body weight

SECONDARY OUTCOMES:
Fidelity of delivery to the intervention | throughout intervention delivery, which can range from 2-4 years for parent educators depending on when their site is randomized
  Parent educators' fidelity to the intervention will all be assessed using a coding document (developed for the current study), which will be applied to audio-recordings of study visits, and will document the following components: adherence, quality of delivery, exposure to the intervention, and participant responsiveness or involvement, all of which share a common unit of measure

CONTACTS AND LOCATIONS:
Overall Officials: Debra Haire-Joshu, PhD, Principal Investigator — Washington University School of Medicine; Rachel G Tabak, PhD, RD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided
Only data with identifiers removed will be shared publicly. Any identified data to be shared will only be done so in coordination with the Human Research Protection Office at Washington University in St. Louis and the Institutional Review Board (IRB) at the requesting investigator's institution.
  Datasets with identifiers will only be accessible to study team members with appropriate Human Subjects training.